CLINICAL TRIAL: NCT02588183
Title: PV Cryoablation Efficacy Using Electrophysiological Endpoints and the New Generation ArticFont Advance ST Catheter (COR ADVANCE Study)
Brief Title: PV Cryoablation Efficacy (COR ADVANCE Study)
Acronym: COR-ADVANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Nicasio Perez Castellano, FEA, Hospital San Carlos, Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AF-3064: COR ADVANCE Study
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; pulmonary vein; cryoenergy; cryoablation; ArcticFront
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ArticFont Advance ST (Experimental): Patients undergoing PV isolation with the ArticFont Advance ST Cryoenergy Balloon Catheter
  Interventions: Device: ArticFont Advance ST Cryoenergy Balloon Catheter

INTERVENTIONS:
Device: ArticFont Advance ST Cryoenergy Balloon Catheter — PV isolation using the ArticFont Advance ST Cryoenergy Balloon Catheter

SUMMARY:
The COR advance study is a non-randomized prospective single center study to assess the results of an electrophysiologically guided approach for PV cryoablation using the Arctic Front Advance ST® catheter together with the Achieve® mapping catheter in 25 patients with drug-refractory paroxysmal AF.

Methods Patient selection criteria will be the same that in the original COR study. All patients will be followed with a Reveal LINQ® cardiac monitor that will be implanted before ablation. The primary objective is the proportion of patients remaining free from atrial fibrillation recurrences without taking antiarrhythmic drugs 12 months after ablation. Secondary objectives are: AF-free survival without anti arrhythmic drugs 12 months after ablation, cumulative AF burden (number of AF episodes and percentage of time in AF) 12 months after ablation, percentage of the pulmonary veins with bidirectional block at the end of the procedure, and ablation time (from the onset of the first energy delivery to the end of the last energy delivery), procedure time (from femoral puncture to catheter removal), and fluoroscopy time.

Final results will be known 24 months after the first enrollment. Statistical analysis Continuous variables that are distributed normally according to the Shapiro-Wilk test will be presented as the mean [standard deviation], and the values will be compared with the t test. Continuous variables that do not follow a normal distribution will be presented as the median [25th to 75th percentile] and will be compared with the Mann-Whitney U test. Categorical variables between two groups with expected values <5 will be compared with the Fisher exact test. Otherwise, categorical variables will be compared with the chi-squared test. The AF-free survival functions will be represented as Kaplan-Meier curves. Data analyses will be done with JMP® (version 9.0.1, SAS Institute Inc., Cary, NC, USA) and Stata® (version 11.0, StataCorp LP; College Station, TX, USA).

DETAILED DESCRIPTION:
Background The Cryoenergy Or Radiofrequency [COR] trial is a randomized, single-center study that compared the efficacy of a anatomical simplified strategy for pulmonary vein cryoballoon ablation (2 shots per PV, 1 first-generation Arctic Front® catheter per patient and no additional touch-up applications to close residual gaps) versus the standard technique for pulmonary vein isolation using open-irrigated radiofrequency catheters (Navistar Thermocool®) with electrophysiological (Lasso®) and electroanatomical guidance (Carto 3®) in 50 patients with drug-refractory paroxysmal atrial fibrillation. All patients were followed with an implantable cardiac monitor (Reveal XT®).

The primary endpoint of the study (proportion of patients remaining free from atrial fibrillation recurrences without taking antiarrhythmic drugs 12 months after ablation) was met by 48% of patients treated with cryoenergy and 68% of patients treated with radiofrequency (OR 0.43 [95% confidence interval, 0.19 to 1.0]; P=0.05). This difference disappeared after adjustment for acute procedural outcome. In patients for whom all 4 PVs were blocked at the end of the procedure, there was no difference between group C and group R in the primary endpoint (67% versus 68%; P=0.94). Thus, the COR trial supports that: 1) complete PV conduction block is critical to the success of AF ablation; 2) despite the fact that the results of the anatomical cryoablation technique used in the COR study are superior to the previously published series of patients treated with PV cryoablation and followed by implantable monitors, results of cryoablation might be even better if we aim for PV conduction block. At present time, the availability of the Achieve® mapping catheter and the more efficient 2nd-generation cryoballoon ArcticFront Advance® catheter provides an opportunity to test a electrophysiologically guided PV cryoablation approach against conventional PV isolation with point-by-point radiofrequency ablation catheters.

The COR advance study is a non-randomized observational prospective single center study to assess the results of an electrophysiologically guided approach for PV cryoablation using the Arctic Front Advance ST® catheter together with the Achieve® mapping catheter in 25 patients with drug-refractory paroxysmal AF.

Methods

Inclusion criteria:

* Symptomatic recurrent paroxysmal AF
* >2 episodes in the last 6 months
* Refractory to 1 or more antiarrhythmic drugs
* Anatomical pattern consisting of 4 pulmonary veins
* Willing and capable of providing informed consent

Exclusion criteria:

* Patients that are <18 or >75 years old
* Prior AF ablation
* Prior cardiac surgery
* Moderate to severe valvular heart disease
* Anteroposterior diameter of the left atrium >50 mm
* Hyperthyroidism, intracardiac thrombus, contraindications for anticoagulation, concomitant acute illness, pregnancy.
* Unavailability for follow-up at our center for at least 1 year

All procedures will be performed in the Arrhythmia Unit of our Institution. Patients will need to give written informed consent to be enrolled in this study. Pre-procedural exams and pre-ablation technique will be the same that used in the COR trial. The end point of PV cryoablation will be complete bidirectional PV conduction block assessed with the Achieve® catheter. Only one ArcticFront Advance® or ArcticFront Advance ST® catheter (23 or 28 mm diameter) will be used per patient. Every cryoenergy delivery will last 240 seconds, except in case of excessive freezing (temperature ≤-65ºC with a 23 mm balloon or ≤-60º with a 28 mm balloon), diaphragmatic hypokinesia or other significant adverse event related to freezing. No bonus applications will be given if the time to effect is less than 60 seconds with a 23-mm cryoballoon catheter, or less than 90 seconds with a 28-mm cryoballoon. When the time to effect cannot be assessed, no bonus applications will be given provided that there is complete occlusion of the PV during freezing (persistent contrast staining of the PV) and the application results in PV conduction block. Otherwise, either late PV conduction block or incomplete PV occlusion during freezing will need a bonus cryoenergy delivery. If PV conduction block is not achieved, one or more additional cryoenergy applications will be given at discretion of the responsible physician. Thus, the number of cryoenergy applications will not be limited by protocol, but the use of a different size cryoballoon or conventional point-by-point ablation catheters is strongly discouraged.

Patient selection criteria will be the same that in the original COR study. All patients will be followed with a Reveal LINQ® cardiac monitor that will be implanted before ablation. The primary objective is the proportion of patients remaining free from atrial fibrillation recurrences without taking antiarrhythmic drugs 12 months after ablation. Secondary objectives are: AF-free survival without anti arrhythmic drugs 12 months after ablation, cumulative AF burden (number of AF episodes and percentage of time in AF) 12 months after ablation, percentage of the pulmonary veins with bidirectional block at the end of the procedure, and ablation time (from the onset of the first energy delivery to the end of the last energy delivery), procedure time (from femoral puncture to catheter removal), and fluoroscopy time.

Final results will be known 24 months after the first enrollment.

Statistical analysis Continuous variables that are distributed normally according to the Shapiro-Wilk test will be presented as the mean [standard deviation], and the values will be compared with the t test. Continuous variables that do not follow a normal distribution will be presented as the median [25th to 75th percentile] and will be compared with the Mann-Whitney U test. Categorical variables between two groups with expected values <5 will be compared with the Fisher exact test. Otherwise, categorical variables will be compared with the chi-squared test. The AF-free survival functions will be represented as Kaplan-Meier curves. Data analyses will be done with JMP® (version 9.0.1, SAS Institute Inc., Cary, NC, USA) and Stata® (version 11.0, StataCorp LP; College Station, TX, USA).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic recurrent paroxysmal AF
* >2 episodes in the last 6 months
* Refractory to 1 or more antiarrhythmic drugs
* Anatomical pattern consisting of 4 pulmonary veins
* Willing and capable of providing informed consent

Exclusion Criteria:

* Patients that are <18 or >75 years old
* Prior AF ablation
* Prior cardiac surgery
* Moderate to severe valvular heart disease
* Anteroposterior diameter of the left atrium >50 mm
* Hyperthyroidism, intracardiac thrombus, contraindications for anticoagulation, concomitant acute illness, pregnancy.
* Unavailability for follow-up at our center for at least 1 year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08; Primary Completion 2017-03 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients free-from AF, without antiarrhythmic drug therapy | 12 months

SECONDARY OUTCOMES:
AF-free survival, without antiarrhythmic drug therapy | 12 months
Proportion of PV with bidirectional block | intraoperative
Time required to complete isolation (LA time) | intraoperative
Cumulative AF burden | 12 months
  Percentage of time in AF (%) and number of AF episodes (n)

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Arritmias, Hospital Clínico San Carlos, Madrid, Spain

REFERENCES:
- [Result] Perez-Castellano N, Fernandez-Cavazos R, Moreno J, Canadas V, Conde A, Gonzalez-Ferrer JJ, Macaya C, Perez-Villacastin J. The COR trial: a randomized study with continuous rhythm monitoring to compare the efficacy of cryoenergy and radiofrequency for pulmonary vein isolation. Heart Rhythm. 2014 Jan;11(1):8-14. doi: 10.1016/j.hrthm.2013.10.014. Epub 2013 Oct 5. PMID 24103221